CLINICAL TRIAL: NCT02696330
Title: Comparison Between Effect of Enoxaparin and Clopidogrel on Improving Pregnancy Rate in ICSI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Amr Ahmed Mahmoud Riad, Lecturer of obstetrics and gynecology, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICSI
Record Dates: First submitted 2016-02-12; First posted 2016-03-02 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Female , Infertility
MeSH Terms: conditions — Infertility, Female | interventions — Clopidogrel; Enoxaparin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- clopidogrel (Active Comparator): 50 patients undergoing ICSI
  Interventions: Drug: clopidogrel
- enoxaparin (Active Comparator): 50 patients undergoing ICSI
  Interventions: Drug: enoxaparin
- placebo (Placebo Comparator): 50 patients undergoing ICSI
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: clopidogrel — clopidogrel 75mg tablets with 300mg loading dose followed by 75mg oral tablets daily starting from day of hCG trigger till assessment of pregnancy by ultrasound
  Other Names: plavix
  Arms: clopidogrel
Drug: enoxaparin — enoxaparin 40 mg by subcutaneous injection once daily starting from day of hCG trigger till assessment of pregnancy by ultrasound
  Other Names: clexane
  Arms: enoxaparin
Drug: placebo — starch tablets with no active drug material is given daily starting from day of hCG trigger till assessment of pregnancy by ultrasound
  Arms: placebo

SUMMARY:
Comparison between effect of enoxaparin and clopidogrel on improving pregnancy rate in ICSI

DETAILED DESCRIPTION:
Study setting:

Assisted Reproduction unit in Ain Shams University Maternity Hospital

Study population:

Patients underlying ICSI in Assisted Reproduction unit in Ain Shams University maternity hospital

Intervention:

After taking written informed consent, all patients recruited in the study will undergo, detailed medical history and complete clinical examination will be obtained along with necessary laboratory investigations and ultrasound findings The standard protocol of the Assisted Reproduction unit in Ain Shams University Maternity Hospital for induction of ovulation in ICSI patients which it is the long protocol will be given for all patients in the study. Endometrial and sub-endometrial blood flow for every patient in the 3 groups will be assessed by transvaginal ultrasound using Medison Sonoace R5 ultrasound machine, eight hours before giving the trigger, after they have completely emptied their bladders (2D power Doppler will be performed). This will be repeated one week after the day of embryo transfer. Endometrial blood flow will be detected by intra-endometrial or the adjacent sub-endometrial regions within 10 mm of the echogenic endometrial borders. Double thickness of the endometrium will be measured (maximum distance between each myometrial/endometrial interface through the longitudinal axis of the uterus). The pulsatility index (PI) and resistance index (RI) of the endometrial arteries will be calculated. Analysis will be used together with computer algorithms to form indices of blood flow within the endometrium. The parameters will be analyzed by software for: (i) resistance index (RI): the difference between maximal systolic blood flow and minimal diastolic flow divided by the peak systolic flow (S-D/S); (ii) pulsatility index (PI): the difference between maximal systolic blood flow and minimal diastolic flow divided by the mean flow throughout the cycle (S - D/mean); (iii) the ratio between peak systolic flow and lowest diastolic flow (S/D). These three parameters express the resistance to flow from the point of measurement downstream. The patients will be divided into three groups according to the condition of the endometrial blood flow: In Group 1, no endometrial blood flow is detected; Group 2 has sub-endometrial blood flow detected, and Group 3 has both endometrial and sub-endometrial blood flow detected.

Pregnancy will be assessed by serum B-HCG test after fourteen days of having embryo transfer, then two weeks later trans-vaginal ultrasound will be performed to insure the presence of gestational sac.

ELIGIBILITY:
Inclusion Criteria:

Age :20-35yrs.

1. Embryo transfer at 3rd or 5th day after ovum pick up.
2. The transferred embryos are in the four cell stage ,eight cell stage, sixteen cell stage or blastocyst stage.

Exclusion Criteria:

1. Age <20 or >35 yrs old.
2. Chronic medical disease.
3. Single embryo transfer.
4. Previous ICSI failure.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy | 24 hours
  number of participants with positive serum hCG indicating pregnancy

SECONDARY OUTCOMES:
endometrial and subendometrial blood flow | 24 hours
  number of participants with improved endometrial and subendometrial blood flow by 2D Doppler ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams maternity hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided